CLINICAL TRIAL: NCT04596618
Title: Impact of Forearm Immersion Cooling Equipment (ICE) on Exercise Performance in the Heat
Brief Title: Impact of ICE on Exercise Performance in the Heat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Douglas J Casa, Professor, University of Connecticut
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H20-0092
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Participants receive two cooling treatments on separate study visits: 1) passive cooling 2) forearm immersion cooling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forearm Cooling (Active Comparator): Participants will be actively cooled during rest breaks.
  Interventions: Device: Forearm cooling
- No Forearm Cooling (No Intervention): Participants will participant in "passive cooling" where they sit in a chair during rest.

INTERVENTIONS:
Device: Forearm cooling — forearm cooling will be performed for active cooling assessment.
  Arms: Forearm Cooling

SUMMARY:
The purpose of this study is to determine the effects of intermittent forearm cooling on exercise performance in the heat.

DETAILED DESCRIPTION:
The study will be completed in the following timeline:

Visit 1: Baseline and VO2max testing. Visit 2-3: Trial 1 and 2

Visit specific information is described below, however, specific data collection protocols for dependent variables and procedures are included below the description of the study design.

Visit 1: Baseline and VO2max Testing

Participants who are approved to participate will be scheduled for a baseline and VO2max testing day. Upon arrival to the lab, subjects will provide a urine sample in a clean urine cup. Urine specific gravity and urine color will be assessed. Nude body mass will be also be recorded. Privacy will be afforded for each participant while obtaining body mass measures by taking measurements with the participant alone in a private room behind a solid, closed door, and the research reading the scale outside of the room. Participants will only be permitted to continue to the VO2max test if the euhydrated criteria of a urine specific gravity (USG) <1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. Height will be measured with a tape measure on Visit 1. Percent body fat will be calculated using a 3-site evaluation of skin fold thickness using skin fold calipers. A researcher will use appropriate grasping technique to measure skin fold thickness on the chest, tricep, and abdomen. This will take less than 5 minutes to complete. This information will be used to describe the subject demographics. Participants will also be asked to complete a maximal oxygen uptake (VO2max) test on a treadmill in a thermoneutral environment. This test will provide aerobic fitness levels of the participants. This visit will take approximately 1-2 hours.

Visit 2-3: Trials 1 and 2

Participant numbers will be randomly assigned, and trials will be ordered with a random number generator and assigned to a participant number. These orders will be counterbalanced between participants to ensure that there is not an order effect, and each participant will complete two trials as part of the study. Participants will be allowed to make-up trial visits if they are sick, suffer an injury or do not meet hydration requirements. Participants will be asked if they have a current illness or taking medications to determine whether they can complete the exercise trial. The participant's visit will be rescheduled if they have a fever, current illness or taking medications that influence body temperature.

Participants will complete two trials on two separate days in a randomized counter balanced order:

Trial Cooling Intervention

1. Passive Cooling
2. Forearm Immersion

The exercise protocol, cooling intervention, and performance battery portions of this study will be conducted in a climatic chamber with ambient temperature approximately 30-40C and relative humidity at approximately 40-60%. Participants will drink approximately 1.4L of water throughout the exercise trial. Upon arrival to the lab, participants will be asked to indicate if they have consumed alcohol or caffeine in the last 24 hours and 12 hours, respectively. They will not be asked to specify exactly what they have consumed, but if they provide a positive indication, their trial will be rescheduled for another day. Participants will provide a small urine sample in a clean urine cup, and a nude body mass will be measured. Upon arrival to the lab, hydration status will be assessed by urine specific gravity, nude body mass and urine color. Participants will only be permitted to continue to the exercise trial if the euhydrated criteria of a urine specific gravity (USG) <1.025 is met. If the participant arrives with a USG between 1.020 and 1.025, the subject will be asked to drink 500 mL of water to ensure proper hydration status. Participants will be given instructions at the prior visit about how to obtain desired hydration status for the upcoming trial. Participants will insert a rectal probe and wear a heart rate monitor strap. Researchers will insert the esophageal probe. Additionally, participants will wear 4-site skin temperature sensors. Researchers will apply the skin temperature sensors with medical tape to the participants' chest, upper arm, thigh, and calf.

Participants will enter the environmental chamber and sit for 10 minutes to become equilibrated. Participants will wear a metabolic mask during this time to assess baseline metabolic heat production. The environmental chamber will be set to 35C ambient temperature, 50% relative humidity. After baseline measures of heart rate, rectal temperature, and metabolic heat production, participants will complete the perceptual indices. Participants will also complete an environmental symptoms questionnaire (ESQ).

The trial will consist of three, 20-minute exercise bouts consisting of walking, running, and sprinting at varying speeds ranging approximately 20-90% of their VO2max. Followed by a 12-minute "half-time" consisting of passive rest. Participants will then complete three more 20-minute exercise bouts consisting of walking, running, and sprinting at varying speeds ranging approximately 20-90% of their VO2max, for a total of six 20-minute bouts.

Each 20-minute exercise bout with be followed by a 3-minute break where cooling will occur. Participants will be allowed to drink 750mL of water throughout each exercise half for a total of 1.4L. The participant will be cooled for approximately 3 minutes after each 20-minute exercise bout with their assigned cooling modality. Rectal temperature, esophageal temperature, skin temperature, heart rate, perceptual measures, and metabolic heat production will be collected at various time points before, during, and after exercise and cooling. Following the completion of the six 20-minute exercise bouts, participants will perform the performance battery. The performance battery will consist of an agility test, grip strength test, broad-jump test, sprint test, and 1-mile time trial test.

Passive Cooling: Participants will be asked to sit in a chair in the climate chamber for passive cooling.

Forearm immersion: The participant will place both of their forearms in approximately 15C water during forearm immersion.

Each trial will be approximately 3 hours.

All devices will be properly cleaned according to manufacturer's instruction prior to use by other participants.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender male between the ages of 18-30 years
* been cleared by the medical monitor for the study
* VO2max >45ml/kg/min

Exclusion Criteria:

* 1. have a current musculoskeletal injury that would limit their physical activity or preclude the participant from walking, jogging, running, sprinting, or cutting.

  2. Chronic health problems that affect your ability to thermoregulate (disorders affecting the liver, kidneys or the ability to sweat normally) 3. Fever or current illness at the time of testing 4. History of cardiovascular, metabolic, or respiratory disease 5. Current musculoskeletal injury that limits their physical activity 6. Currently taking a medication that is known to influence body temperature (amphetamines, antihypertensives, anticholinergics, acetaminophen, NSAIDs, aspirin) 7. Are a female 8. Have a history of heat related illness 9. Have any cold allergies or adverse reactions to the cold (i.e. cold urticaria, Raynaud's, cryoglobulinemia)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Change in Rectal Temperature | Measured continuously during the duration of the trial (total 150 minutes)
  Rectal thermometer will be self-inserted by participant to assess core temperature
Change in Mean Skin Temperature | Measured continuously during the duration of the trial (total 150 minutes)
  4 skin temperature sensors will be placed on the subject (chest, shoulder, thigh, calf)
Change in Heart Rate | Measured continuously during the duration of the trial (total 150 minutes)
  A heart rate monitor will be worn by participant throughout exercise/cooling protocol
Change in Esophageal Temperature | Measured continuously during the duration of the trial (total 150 minutes)
  An esophageal thermometer will be inserted by the researchers to assess participants esophageal temperature.
Change in Rating of Perceived Exertion (RPE) | Measured every 5 minutes during the duration of the trial (total 150 minutes)
  6-20 scale that indicates how hard the participant feels they are working. 6 represents rest and 20 represents maximal exertion. A high score indicates more perceived exertion.
Change in Thermal Sensation (TS) | Measured every 5 minutes during the duration of the trial (total 150 minutes)
  0-8 Scale (cold to hot) that indicated how cold or hot the participate feels. 0 = extremely cold, 8 = extremely hot.
Change in Perception of Fatigue | Measured every 5 minutes during the duration of the trial (total 150 minutes)
  0-10 (no fatigue to extreme fatigue) Scale that indicates how fatigued the participate feels. High score indicates more fatigue (negative outcome).
Change in Perception of Thirst | Measured every 5 minutes during the duration of the trial (total 150 minutes)
  0-9 (no thirst to extreme thirst) Scale that indicates how thirsty the subject feels. A higher score is considered a negative outcome.
Environmental Symptoms | Before the start of exercise block 1
  An environmental symptoms questionnaire to indicate they feel (hot, lethargic, irritable) with the scale ranging from Not at all, a little, somewhat, moderate, a lot, to extreme.
Environmental Symptoms | After completion of the performance battery, at time point 180min.
  An environmental symptoms questionnaire to indicate they feel (hot, lethargic, irritable) with the scale ranging from Not at all, a little, somewhat, moderate, a lot, to extreme.
Quick-Board Agility | After the end of 3min cooling period block 6
  Agility will be assessed by number of foot taps within 10seconds and then number of hops within 10seconds.
Broad Jump | after the quick-board agility, at time point 153minutes
  Participants will attempt to jump as far forward as they can 3 times, measured in centimeters.
Grip Strength | after the Broad jump test, at time point 155minutes
  Participants will squeeze a hand held dynamometer 3 times, measured in kilograms
Sprints | after the grip strength test, at time point 160minutes
  On a non-motorized treadmill, participants will sprint for 6sec followed by 24sec of rest, repeat 3 times, belt revolutions will be measured.
One Mile Timed Trial | after the sprint test, at time point 170minutes
  On a motorized treadmill, participants will run at a self-selected pace until they run a distance of 1-mile, time measured in minutes
Metabolic heat production | Measured during the last 5 minutes of each exercise block for a total of six measurements for a total of 36minutes.
  Using a metabolic mask and metabolic cart, metabolic heat production will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Casa, PhD, Principal Investigator — University of Connecticut
Locations (1):
- Gampel Pavilion, Storrs, Connecticut, United States